CLINICAL TRIAL: NCT00355862
Title: A Prospective Randomised, Open-labeled, Trial Comparing Sirolimus-Containing Versus mTOR-Inhibitor-Free Immunosuppression in Patients Undergoing Liver Transplantation for Hepatocellular Carcinoma
Brief Title: Immunosuppression in Patients Undergoing Liver Transplantation for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Edward K Geissler, Regensburg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SiLVER05; EudraCT Number:; 2005-005362-36
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Sirolimus; mTOR; HCC-recurrence free survival; Liver transplant recipients; HCC recurrence free survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cni protein, Drosophila; Steroids; Cyclosporine; Tacrolimus; Azathioprine; Prednisolone; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Center specific immunosuppressive regimen (mTOR inhibitor free)
  Interventions: Drug: CNI, MMF, Steroids, Aza etc. (mTOR inhibitor free)
- 2 (Experimental): Sirolimus containing regimen
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: CNI, MMF, Steroids, Aza etc. (mTOR inhibitor free) — center specific therapeutic regimen without mTOR inhibition
  Other Names: Cyclosporine; Tacrolimus; Azathioprine; MMF; Prednisolone; etc
  Arms: 1
Drug: Sirolimus — Sirolimus based immunosuppression
  Other Names: Rapamune
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of sirolimus-based immunosuppressive therapy in patients following orthotopic liver transplantation (OLT) for hepatocellular carcinoma (HCC), with regard to HCC recurrence-free patient survival.

DETAILED DESCRIPTION:
There are two major issues to face in patients who underwent liver transplantation for hepatocellular carcinoma (HCC). First, the patient requires adequate immunosuppressive medication to avoid rejection of its allograft. Second, the risk for HCC recurrence has to be reduced to a minimum.

To date, it is a wide spread argument that immunosuppressive agents for the reduction of allograft rejection are generally tumorogenic, or at least are permissive of cancer development although little is known about their tumorogenic effect. In clinical studies substantiated by experimental data, cyclosporin (CsA) enhances cancer cell growth characteristics and angiogenesis in tumors and inhibits DNA repair mechanisms, promoting their growth. In an experimental rat-model CsA promoted liver tumor recurrence and growth. In other experimental studies a higher proliferation rate of human hepatoma cells in the presence of tacrolimus was demonstrated.

Nevertheless not all immunosuppressive agents do necessarily promote tumor growth, and in fact, can have antineoplastic activities. Sirolimus, in immunosuppressive doses, has potent antiangiogenic properties that inhibit tumor growth. The antiangiogenetic mechanism is due to inhibition of vascular endothelial growth factor (VEGF) production and signaling to endothelial cells. Besides that, sirolimus directly blocks critical intracellular pathways (mTOR) and inhibits cell-cycle. Through increased E-cadherin expression on tumor cells, tumor metastasis can be reduced by increased tumor cell binding.

In this context it has to be mentioned that in mouse models where a transplant recipient also has a tumor, the pro-tumor effects of CsA are completely negated by sirolimus.

Especially HCC seems to be particularly sensitive to VEGF/angiogenesis, indicating a potential susceptibility to the action of sirolimus which could be shown by the group of E.K. Geissler and colleagues in Regensburg.

From a clinical perspective there is a recent pilot study from Kneteman et al. indicating that early conversion of immunosuppression from CNI to mTOR-inhibitors after OLT in HCC patients (n=21) with a "high risk" for tumor recurrence results in a tumor recurrence rate of only 19% and a 4-year over all survival of 83% in this group. Moreover, in the "low-risk" group (n=19) the 4-year tumor recurrence rate was only 1/19. Post-HCC recurrence survival was 15.5 months, which is marked improvement compared to currently published data. Although this study only reports on a small number of patients and is not controlled, it suggests the potential role for sirolimus to ameliorate tumor recurrence, leading to a more benign course of renewed tumor disease.

Among the most serious complications of immunosuppressive therapy in organ transplantation is the high risk of previous neoplasia recurrence, or the development of de novo cancer. HCC comprises 80-90 % of malignancies indicating OLT. Before the introduction of strict criteria for the enrollment of primary liver tumors, tumor recurrence led to poor mid- and long-term results. HCC thus has an unacceptable recurrence rate following OLT when the tumor exceeds 5 cm in size. ELTR data from 2003 showed a 5 year patient overall survival for hepatic malignancy (including more than 80% HCC in this group since 1997) of merely 53%, comparing poorly with data from non-cholestatic liver cirrhosis of 74% and even acute liver failure of 62%. Based on previous work, and a landmark publication in 1996 by Mazzaferro et al. many centers have restricted their indication for liver transplantation due to clinical criteria based on tumor size and number to the so-called ´Milan Criteria´.

Implementing these criteria, recent single center data show an improvement in both disease-free and overall survival following OLT for HCC. Nevertheless approximately 30% of patients in these studies who were thought to be within Milan Criteria before transplantation, proved by histopathological examination to have extended disease. This led to a dramatic decline in overall and disease-free survival, from 71-85% to 40-50%, and from 65-78% to 27-30%, respectively.

In total all preclinical and clinical observations have led us to the purpose that the use of sirolimus in HCC patients could improve survival after liver transplantation by decreasing tumor recurrence rate. Thus patients should experience less posttransplant problems with HCC recurrence, and therefore could expect a longer, and better quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Histologically proven HCC before randomisation
3. Signed, written informed consent

Exclusion Criteria:

1. Multiple-organ recipients.
2. Known hypersensitivity to sirolimus or its derivatives.
3. Hyperlipidemia refractory to optimal medical management. (cholesterol >300 mg/dL; triglycerides >350 mg/dL).*
4. Evidence of significant local or systemic infection.
5. Known HIV-positive patients.*
6. Platelets <75,000/cubic mm.*
7. Women of child-bearing potential not willing to take contraception.
8. Patients with non-HCC malignancies within the past 5 years,excluding successfully treated squamous cell carcinoma and basal cell carcinoma of the skin.
9. Extrahepatic HCC tumor manifestation
10. Patients with a psychologic, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule.
11. Patients under guardianship (e.g. individuals who are not able to freely give their informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | 5 year follow up after last patient in

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Geissler, Prof. PhD, Study Chair — Regensburg University Medical Center, Head of Experimental Surgery; Hans J Schlitt, Prof. MD. FACS FRACS FRCS MHM, Study Director — Regensburg University Medical Center, Director of Surgical Department; Andreas A Schnitzbauer, MD, Principal Investigator — Regensburg University Hospital
Locations (1):
- Regensburg University, Regensburg, Bavaria, Germany

REFERENCES:
- [Derived] Schnitzbauer AA, Filmann N, Adam R, Bachellier P, Bechstein WO, Becker T, Bhoori S, Bilbao I, Brockmann J, Burra P, Chazoullieres O, Cillo U, Colledan M, Duvoux C, Ganten TM, Gugenheim J, Heise M, van Hoek B, Jamieson N, de Jong KP, Klein CG, Klempnauer J, Kneteman N, Lerut J, Makisalo H, Mazzaferro V, Mirza DF, Nadalin S, Neuhaus P, Pageaux GP, Pinna AD, Pirenne J, Pratschke J, Powel J, Rentsch M, Rizell M, Rossi G, Rostaing L, Roy A, Scholz T, Settmacher U, Soliman T, Strasser S, Soderdahl G, Troisi RI, Turrion VS, Schlitt HJ, Geissler EK. mTOR Inhibition Is Most Beneficial After Liver Transplantation for Hepatocellular Carcinoma in Patients With Active Tumors. Ann Surg. 2020 Nov;272(5):855-862. doi: 10.1097/SLA.0000000000004280. PMID 32889867
- [Derived] Geissler EK, Schnitzbauer AA, Zulke C, Lamby PE, Proneth A, Duvoux C, Burra P, Jauch KW, Rentsch M, Ganten TM, Schmidt J, Settmacher U, Heise M, Rossi G, Cillo U, Kneteman N, Adam R, van Hoek B, Bachellier P, Wolf P, Rostaing L, Bechstein WO, Rizell M, Powell J, Hidalgo E, Gugenheim J, Wolters H, Brockmann J, Roy A, Mutzbauer I, Schlitt A, Beckebaum S, Graeb C, Nadalin S, Valente U, Turrion VS, Jamieson N, Scholz T, Colledan M, Fandrich F, Becker T, Soderdahl G, Chazouilleres O, Makisalo H, Pageaux GP, Steininger R, Soliman T, de Jong KP, Pirenne J, Margreiter R, Pratschke J, Pinna AD, Hauss J, Schreiber S, Strasser S, Klempnauer J, Troisi RI, Bhoori S, Lerut J, Bilbao I, Klein CG, Konigsrainer A, Mirza DF, Otto G, Mazzaferro V, Neuhaus P, Schlitt HJ. Sirolimus Use in Liver Transplant Recipients With Hepatocellular Carcinoma: A Randomized, Multicenter, Open-Label Phase 3 Trial. Transplantation. 2016 Jan;100(1):116-25. doi: 10.1097/TP.0000000000000965. PMID 26555945
- [Derived] Schnitzbauer AA, Zuelke C, Graeb C, Rochon J, Bilbao I, Burra P, de Jong KP, Duvoux C, Kneteman NM, Adam R, Bechstein WO, Becker T, Beckebaum S, Chazouilleres O, Cillo U, Colledan M, Fandrich F, Gugenheim J, Hauss JP, Heise M, Hidalgo E, Jamieson N, Konigsrainer A, Lamby PE, Lerut JP, Makisalo H, Margreiter R, Mazzaferro V, Mutzbauer I, Otto G, Pageaux GP, Pinna AD, Pirenne J, Rizell M, Rossi G, Rostaing L, Roy A, Turrion VS, Schmidt J, Troisi RI, van Hoek B, Valente U, Wolf P, Wolters H, Mirza DF, Scholz T, Steininger R, Soderdahl G, Strasser SI, Jauch KW, Neuhaus P, Schlitt HJ, Geissler EK. A prospective randomised, open-labeled, trial comparing sirolimus-containing versus mTOR-inhibitor-free immunosuppression in patients undergoing liver transplantation for hepatocellular carcinoma. BMC Cancer. 2010 May 11;10:190. doi: 10.1186/1471-2407-10-190. PMID 20459775
- [Derived] Geissler EK. Rapamycin enhances lifespan: at last, an advantage for transplant recipients? Nephrol Dial Transplant. 2009 Dec;24(12):3623-5. doi: 10.1093/ndt/gfp496. Epub 2009 Sep 22. No abstract available. PMID 19773418
- [Derived] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962
- See also: Related Info — http://www.klinikum-regensburg.de